CLINICAL TRIAL: NCT00442169
Title: Randomized, Double-blind, Placebo Controlled Phase II Trial of the Safety, Tolerability and Immunogenicity of Lyophilized ChimeriVax-WN02 West Nile Vaccine in Healthy Adults
Brief Title: Safety and Immunogenicity of ChimeriVax-WN02 West Nile Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-244-003
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: West Nile Fever
Keywords: West Nile Disease; Antibody response; Viremia; Safety; Tolerability; Prevention
MeSH Terms: conditions — West Nile Fever; Viremia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: WN02 Low Dose (Part 1) (Experimental): Low Dose in healthy adults in Part 1 against a placebo control.
  Interventions: Biological: ChimeriVax-WN02 Low Dose
- Group 2: WN02 Medium Dose (Part 1) (Experimental): Medium dose level in part one healthy subjects against a placebo control.
  Interventions: Biological: ChimeriVax-WN02 Medium Dose
- Group 3: WN02 High Dose (Part 1) (Experimental): High dose level in part one healthy subjects against a placebo control
  Interventions: Biological: ChimeriVax-WN02 High Dose
- Group 4: Placebo (Part 1) (Placebo Comparator): Participants will receive a single dose of saline in Part 1 on Day 0
  Interventions: Biological: 0.9% Saline solution
- Group 5: WNO2 High Dose (Part 2) (Experimental): Participants enrolled in Part 2 and received a single dose of West Nile Virus vaccine.
  Interventions: Biological: ChimeriVax-WN02 High Dose
- Group 6: Placebo (part 2) (Placebo Comparator): Participants will receive a single dose of saline in Part 2 on Day 0
  Interventions: Biological: 0.9 % NaCl solution

INTERVENTIONS:
Biological: ChimeriVax-WN02 Low Dose — Single dose formulation given in a volume of 0.5 mL by subcutaneous injection to the deltoid region.
  Arms: Group 1: WN02 Low Dose (Part 1)
Biological: ChimeriVax-WN02 Medium Dose — Single dose formulation given in a volume of 0.5 mL by subcutaneous injection to the deltoid region
  Arms: Group 2: WN02 Medium Dose (Part 1)
Biological: ChimeriVax-WN02 High Dose — Single dose formulation given in a volume of 0.5 mL by subcutaneous injection to the deltoid region
  Arms: Group 3: WN02 High Dose (Part 1)
Biological: 0.9% Saline solution — Single dose formulation given in a volume of 0.5 mL by subcutaneous injection to the deltoid region
  Arms: Group 4: Placebo (Part 1)
Biological: ChimeriVax-WN02 High Dose — Single dose formulation given in a volume of 0.5 mL by subcutaneous injection to the deltoid region
  Arms: Group 5: WNO2 High Dose (Part 2)
Biological: 0.9 % NaCl solution — Single dose given in a volume of 0.5 mL by subcutaneous injection to the deltoid region
  Arms: Group 6: Placebo (part 2)

SUMMARY:
The purpose of this study is to determine whether a single subcutaneous injection of ChimeriVax-WN02 vaccine is well tolerated, safe and induces protective antibodies against West Nile Disease. The study is divided into two parts; in the first part, a comparison of 3 dose levels of the vaccine will be made, with an inactive control. In the second part, the optimum dose level chosen after the first part will be given to older volunteers.

DETAILED DESCRIPTION:
West Nile Disease has been carried across the United States by migrating birds since it was first identified in New York city in 1999. It is transmitted by mosquitoes from birds to humans and can cause severe disease in some individuals. There is no specific treatment for West Nile Disease. The target population for a West Nile vaccine is older people, as they are more susceptible to severe disease. This trial includes a dose-finding part with a placebo control in young healthy adults, followed by a placebo-controlled examination of the chosen dose in older healthy adults.

Outcome measures include a comparison of adverse events between active treatment and placebo, a comparison of antibody and viremia measurements between dose levels and across age groups for the dose chosen for Part 2.

ELIGIBILITY:
Inclusion Criteria: Part 1

* Healthy adult aged 18 to 40 years.
* Women of child-bearing potential should be using hormonal contraception.
* Subject had to be available for the study duration, including all planned follow-up visits.

Exclusion Criteria: Part 1

* Previous vaccination against yellow fever or Japanese encephalitis
* History of flavivirus infection
* Any abnormalities of immune system, or using drugs that affect the immune system.
* History of anaphylaxis to foods, bee stings, vaccines or drugs.
* Receipt of blood or blood products within the preceding 6 months.
* Receipt of any vaccine in the preceding 30 days
* Seropositive to hepatitis C virus (HCV), hepatitis B surface antigen (HBsAg) or Human immunodeficiency virus (HIV)
* Lactation or intended pregnancy in female subjects
* Previous or current military service with overseas deployment
* Travel to Mexico or other flavivirus endemic areas in the tropics for periods of four weeks or more in the previous ten years.

Inclusion Criteria: Part 2

* Aged ≥ 41 years.
* Subjects had to be in general good health.
* Unimpaired cognitive performance as assessed by clock drawing test score
* Subject had to be available for all required study visits, including all planned follow-up visits.
* Women of child-bearing potential should be using hormonal contraception.

Exclusion Criteria: Part 2

* Clinically significant abnormalities on the Screening 12-lead electrocardiogram (ECG).
* An acute or chronic medical condition that, in the opinion of the Investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions included, but were not limited to:

  * History of renal impairment
  * History of significant liver disease or hepatic impairment
  * History of diabetes mellitus (except controlled with diet)
  * An arteriosclerotic event during the 6 months prior to enrollment (including but not limited to myocardial infarction or unstable angina, peripheral bypass surgery for revascularization of an extremity, and transient ischemic attack or stroke)
  * Signs of congestive heart failure at the time of enrollment
  * Angina
* Subjects with 3 or more of the following:

  * Age over 50 years
  * Hypercholesterolemia, or significantly abnormal lipid profile, based on medical history
  * Any prior history of cardiovascular disease
  * Significant family history of cardiovascular disease in any immediate relative
  * History of significant collagen vascular disease.
* The unexplained presence of any of the following findings:

  * Any significant episodes of confusion, memory loss, language impairment, other cognitive impairment, or other abnormal behavior if relatively abrupt in onset
  * Clinically significant depression
  * Sudden visual impairment (e.g., loss of vision, double vision)
  * Slurred or abnormal speech
  * Sudden onset of vertigo
  * Focal weakness in any extremity
  * Focal sensory loss in any extremity
  * Impaired balance
  * Impaired gait.
* Subjects with any diagnosis of dementia or associated concomitant medications (e.g., Aricept) used for treating dementia.
* Subjects with active or a history of neurologic disease or injury, including, but not limited to: Parkinson's, Guillain Barre, epilepsy (except febrile seizures in youth not treated with medication), cerebrovascular accident, head trauma, or any other neurologic condition thought to impact the integrity of the blood-brain barrier.
* Subjects taking warfarin, heparin, or with known bleeding disorders.
* Relative or employee of the study site staff, CRO, or Sponsor participating in this trial.
* A history of vaccination against yellow fever (YF) or Japanese encephalitis. Previous vaccination was determined by history (interview of subject) and/or by reviewing the subject's vaccination card or other official documentation.
* History of flavivirus infection (e.g. West Nile [WN], Systemic Lupus Erythematosus [SLE], Japanese encephalitis, dengue fever).
* History of thymoma, thymic surgery (removal), or myasthenia gravis.
* Known or suspected immunodeficiency disorder, including leukemia, lymphoma, generalized malignancy, or treatment with immunosuppressive medications, including corticosteroids, alkylating agents, anti-metabolites, or radiation therapy. Low dose steroids (≤ 10 mg prednisone or equivalent, topical or intra articular/bursal/tendon/epidural injections of corticosteroids) did not constitute a reason for exclusion.
* History of residence in or travel to Mexico or flavivirus endemic areas in the tropics (India, southeast Asia, Central America, Caribbean, or South America) for periods of 4 weeks or more within the last 10 years.
* Subjects with clinically significant screening laboratory abnormalities and/or those having any of the following:

  * Compromised hematopoietic function defined as a hemoglobin < 10.9 (males) or 9.4 (females) g/dL; lymphocyte count > 3000 mm3; neutrophil count < 1000 mm3; or platelet count < 100,000 mm3.
  * Hepatic dysfunction defined as a bilirubin above upper limit of normal or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 x upper limit of normal.
* Prior history of anaphylaxis to foods, hymenoptera stings, vaccines, or drugs.
* Transfusion of blood or treatment with any blood product, including intramuscular or intravenous serum globulin within 6 months of the Screening Visit or anticipated up to Day 28, or intention to donate blood in the 28 days after vaccination.
* Administration of another vaccine within 30 days preceding the screening visit or anticipated up to Day 28 (these subjects could be rescheduled for vaccination at a later date).
* Physical examination indicating any clinically significant medical condition.
* Subjects with body temperature >37.8ºC/100.0ºF or acute illness within 3 days prior to vaccination (subject could be rescheduled).
* Intention to travel out of the area prior to the study visit on Day 28, such that required study visits would be missed.
* Seropositive to HCV or HIV or positive for HBsAg.
* Participation in another clinical trial within 60 days of Screening.
* Lactation or intended pregnancy in female subjects.
* History of excessive alcohol consumption, drug abuse, or significant psychiatric illness.
* Intention to increase normal exercise routine, participate in contact sports or strenuous weight lifting, or to initiate vigorous exercise from Screening until after Day 28.
* At the time of study or past military service with overseas deployment within 10 years of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (5):
- United States (5):
  - HOPE Research Institute, Phoenix, Arizona
  - Idaho Infectious Diseases, PLLC, Idaho Falls, Idaho
  - PRA International Clinical Pharmacology Center, Lenexa, Kansas
  - Bio-Kinetic Clinical Applications, Inc., Springfield, Missouri
  - The Glennan Centre for Geriatrics and Gerontologyy, EVMS, Norfolk, Virginia

REFERENCES:
- [Derived] Biedenbender R, Bevilacqua J, Gregg AM, Watson M, Dayan G. Phase II, randomized, double-blind, placebo-controlled, multicenter study to investigate the immunogenicity and safety of a West Nile virus vaccine in healthy adults. J Infect Dis. 2011 Jan 1;203(1):75-84. doi: 10.1093/infdis/jiq003. PMID 21148499
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 09 December 2005 to 27 March 2006 in 5 clinical centers in the US.
Pre-assignment Details: A total of 208 participants (Part 1 = 112; Part 2 = 96) who met the inclusion and exclusion criteria were enrolled, randomized, and vaccinated in the study. Report on Part 1 and Part 2 participants with valid data are presented in this report.
Groups:
- Placebo (Part 1): Participants in Part 1 of the study who received a single dose of saline on Day 0
- WN02 Low Dose (Part 1): Participants in Part 1 of the study who received a single dose of West Nile Virus vaccine WN02, 3700 plaque-forming units, on Day 0
- WN02 Medium Dose (Part 1); WN02 High Dose (Part 1): Participants in Part 1 of the study who received a single dose of West Nile Virus vaccine WN02, 37000 plaque-forming units, on Day 0
- Placebo (Part 2): Participants in Part 2 of the study who received a placebo vaccine on Day 0
- WNO2 High Dose (Part 2): Participants in Part 2 of the study who received a single dose of West Nile Virus vaccine WN02, 37000 plaque-forming units, on Day 0
Period: Part 1
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2)
Started | 17 | 24 | 40 | 31 | 0 (Participants in Part 2 are not the same as those in Part 1) | 0 (Participants in Part 2 are not the same as those in Part 1)
Completed | 17 | 24 | 40 | 31 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2)
Started | 0 (Participants in Part 1 are not the same as those in Part 2) | 0 (Participants in Part 1 are not the same as those in Part 2) | 0 (Participants in Part 1 are not the same as those in Part 2) | 0 (Participants in Part 1 are not the same as those in Part 2) | 25 | 57
Completed | 0 | 0 | 0 | 0 | 25 | 57
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2) | Total
Number analyzed (Participants) | 17 | 24 | 40 | 31 | 25 | 57 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 24 | 40 | 31 | 11 | 29 | 152
  >=65 years | 0 | 0 | 0 | 0 | 14 | 28 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.6 (6.41) | 25.4 (5.62) | 25 (5.43) | 25.1 (6.47) | 61.4 (11.8) | 61.0 (11.3) | 25.7 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 19 | 13 | 22 | 40 | 114
  Male | 9 | 12 | 21 | 18 | 3 | 17 | 80
Region of Enrollment [Number; unit: Participants]
  United States | 17 | 24 | 40 | 31 | 25 | 57 | 194

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fourfold or Greater Post-vaccination Titers (Seroconversion).
Description: Seroconversion was defined as a fourfold or greater rise in titer between pre- and post-immunization samples
Time Frame: Day 28 post-vaccination
Population: Seroconversion was assessed in all participants in the safety population according to the vaccine actually received, As Treat Per-Protocol Population
Measure: Number; unit: Participants
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2)
Number analyzed (Participants) | 17 | 21 | 37 | 28 | 25 | 55
Participants | 0 | 21 | 36 | 27 | 0 | 53

2. Secondary Outcome: Geometric Mean Titers of Neutralizing Antibody Titers Pre- and Post-vaccination.
Time Frame: Days 0, 14, and 28 post-vaccination
Population: Geometric mean titers were assessed according to the vaccine actually received, in the As treat per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2)
Number analyzed (Participants) | 17 | 21 | 37 | 28 | 32 | 64
Titers
  Day 0 | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5 [5.0 to 5.0]
  Day 14 | 5.0 [5.0 to 5.0] | 16.8 [7.2 to 39.5] | 35.7 [18.3 to 69.7] | 26.9 [11.8 to 61.5] | 5.0 [5.0 to 5.0] | 19.2 [11.9 to 31.2]
  Day 28 | 5.0 [5.0 to 5.0] | 1367.3 [711.3 to 2628.5] | 2331.1 [1193.3 to 4554.3] | 3309.3 [1726.9 to 6341.7] | 5.0 [5.0 to 5.0] | 922.4 [519.2 to 1638.5]

3. Other Pre Specified Outcome: Number of Participants With Positive Immunoglobulin M (IgM) Response Post-vaccination in the As Treat Per-Protocol Population
Time Frame: Days 14 and 28 post-vaccination
Population: Immunoglobulin M (IgM) response was assessed in all participants in the safety population according to the vaccine actually received, As Treat Per-Protocol Population
Measure: Number; unit: Participants
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2)
Number analyzed (Participants) | 17 | 21 | 37 | 28 | 25 | 56
Participants
  IgM Positive at Day 14 | 0 | 5 | 22 | 10 | 0 | 26
  IgM Positive at Day 28 | 0 | 20 | 36 | 27 | 0 | 53

4. Primary Outcome: Number of Viremic Participants Post-vaccination
Description: Viremic = detectable level of ≥ 10 plaque-forming units (PFU)/mL
Time Frame: Day 21 post-vaccination
Population: Viremia was assessed in all participants in the safety population according to the vaccine actually received.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2)
Number analyzed (Participants) | 17 | 24 | 40 | 31 | 32 | 64
Participants | 2 | 22 | 36 | 29 | 1 | 55

5. Primary Outcome: Treatment-emergent Adverse Events Reported As Related to Study Treatment in at Least 5% of Participants in Any Active Treatment Group Post-vaccination.
Time Frame: Days 0 to 28 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants according to the vaccine actually received, safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2)
Number analyzed (Participants) | 17 | 24 | 40 | 31 | 32 | 64
Participants
  Fatigue | 4 | 1 | 8 | 2 | 5 | 11
  Headache | 5 | 4 | 5 | 2 | 5 | 11
  Malaise | 2 | 1 | 3 | 2 | 3 | 10
  Feeling Hot | 0 | 1 | 1 | 2 | 5 | 11
  Myalgia | 3 | 1 | 3 | 1 | 5 | 13
  Arthralgia | 0 | 1 | 1 | 0 | 3 | 8
  Nausea | 1 | 1 | 2 | 1 | 2 | 5
  Somnolence | 1 | 1 | 2 | 1 | 0 | 5
  Diarrhoea | 0 | 1 | 1 | 0 | 1 | 3
  Chills | 1 | 1 | 1 | 1 | 0 | 4
  Dizziness | 0 | 0 | 1 | 0 | 1 | 2
  Musculoskeletal stiffness | 0 | 1 | 1 | 0 | 5 | 4
  Injection site pain | 2 | 0 | 1 | 0 | 5 | 4
  Pharyngolaryngeal pain | 2 | 0 | 2 | 1 | 2 | 4
  Injection site erythema | NA — Not collected in Part 1 | NA — Not collected in Part 1 | NA — Not collected in Part 1 | NA — Not collected in Part 1 | 6 | 9
  Injection site induration | NA — Not collected in Part 1 | NA — Not collected in Part 1 | NA — Not collected in Part 1 | NA — Not collected in Part 1 | 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination to up to 6 months, post-vaccination.
Arm/Group | Placebo (Part 1) | WN02 Low Dose (Part 1) | WN02 Medium Dose (Part 1) | WN02 High Dose (Part 1) | Placebo (Part 2) | WNO2 High Dose (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/24 | 0/40 | 1/31 | 0/32 | 3/64
Other Adverse Events (participants affected / at risk) | 14/17 | 16/24 | 28/40 | 22/31 | 25/32 | 54/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part 1) (N=17) | WN02 Low Dose (Part 1) (N=24) | WN02 Medium Dose (Part 1) (N=40) | WN02 High Dose (Part 1) (N=31) | Placebo (Part 2) (N=32) | WNO2 High Dose (Part 2) (N=64)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive plumonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part 1) (N=17) | WN02 Low Dose (Part 1) (N=24) | WN02 Medium Dose (Part 1) (N=40) | WN02 High Dose (Part 1) (N=31) | Placebo (Part 2) (N=32) | WNO2 High Dose (Part 2) (N=64)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 7 (7)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 2 (2) | 7 (7)
Chills (General disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 5 (5)
Fatigue (General disorders) | 4 (4) | 2 (2) | 11 (11) | 4 (4) | 7 (7) | 14 (14)
Feeling Hot (General disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 5 (5)
Malaise (General disorders) | 3 (3) | 1 (1) | 7 (7) | 4 (4) | 6 (6) | 14 (14)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 3 (3) | 3 (3) | 4 (5) | 1 (1) | 2 (2)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 5 (5) | 11 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 3 (3)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 5 (5) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 6 (6) | 1 (1) | 5 (5) | 19 (19)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 4 (4) | 0 (0) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 7 (17) | 9 (9) | 14 (14) | 8 (8) | 9 (9) | 18 (18)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (3) | 4 (4) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 9 (9)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 4 (4)
Injection site pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications